CLINICAL TRIAL: NCT06599047
Title: Regional Adipose Tissue Characteristics in Type II Diabetes
Status: Recruiting | Type: Observational
Sponsor: Concordia University, Montreal (Other)
Collaborators: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Principal Investigator, Sylvia Santosa, Professor, Concordia University, Montreal
Other Study IDs: 90000059
Record Dates: First submitted 2024-09-12; First posted 2024-09-19 (Actual); Last update posted 2024-10-22 (Actual); Status verified 2024-10

CONDITIONS: Obesity and Type 2 Diabetes; Bariatric Patients Undergoing Bariatric Surgery; Adipose Tissue Dysfunction Type 2 Diabetes Mellitus Bariatric Surgery; Adipose Tissue Inflammation
Keywords: obesity; Type 2 diabetes; Bariatric Surgery; Adipose Tissue Characterization; Adipose Tissue Inflammation
MeSH Terms: conditions — Obesity; Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Non-Obese Group (Lean): Healthy participants without obesity
- Bariatric Patients without Diabetes: Participants with obesity undergoing bariatric surgery
- Bariatric surgery patients with diabetes: Participants with diabetes undergoing bariatric surgery

SUMMARY:
Fat tissue in different parts of the body has different characteristics. Several studies have associated abdominal fat to an increased risk for multiple metabolic diseases, such as type 2 diabetes and cardiovascular disease, compared with fat located under the skin at the hips and thighs. However, the investigators do not know how the abdominal fat causes or contributes to the development of these diseases or how the development of these disease may in turn cause or contribute to changes in the fat tissue. The general objective of this study is to understand these mechanisms.

To investigate these questions, the study will recruit 140 participants, both men and women aged 18-65 years. The participants will be divided into three groups: 40 people with obesity, 40 with diabetes, and 60 lean individuals. Participants will be recruited from patients at the CIUSSS du Nord-de-l'Île-de Montréal - Hôpital du Sacré-Coeur de Montréal who are awaiting bariatric or general abdominal surgery, as well as from the general population in the Montreal area.

ELIGIBILITY:
Inclusion Criteria:

* Men, premenopausal and postmenopausal females between 18-65 years
* Anticipating having bariatric surgery (participants with obesity) or general surgery in the abdominal area (normal weight participants) with a duration of less than 1.5 hours.
* BMI 30 kg / m2 (participants with obesity)
* Weight Stable for a minimum of two months prior to the first pre-op visit

Exclusion Criteria:

* Smoking
* Renal impairment defined by creatinine clearance; 60 ml/minute
* Uncontrolled hypothyroidism
* No comorbidity other than diabetes type II Exceptions: controlled hypertension, hypothyroidism controlled, controlled dyslipidemia
* Use prescribed medication that affect our outcomes E.g. Exceptions include metformin, DPP-4 inhibitors, inhibitors of the α-glucosidase, hypotensive with a stable dose for 3 months lipid lowering with a stable dose for 3 months.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The Diabetes and Obese groups will be recruited from patients scheduled to undergo bariatric surgery in Montréal and the lean participants will be recruited from healthy patients scheduled to undergo general surgery.
Sampling Method: Non-Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2016-05-01 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Immune Cell Quantification | 5 years
  Flow Cytometry will be used to quantify immune cells in the fat tissue.
Pre-adipocytes and adipocyte characteristics | 5 years
  Cellular characteristics such as proliferation, differentiation and cellular senescence will measured.
Blood Inflammatory Markers | 5 years
  The inflammatory cytokines (e.g. IL6, TNFα), chemokines (e.g. monocyte chemoattractant protein-1), genomics, and adipokines (e.g. leptin, adiponectin) in blood and adipose tissue via PCR, luminex or ELISA will be measured

CONTACTS AND LOCATIONS:
Locations (1):
- Concordia University (School of Health), Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No